CLINICAL TRIAL: NCT04422691
Title: Bruk av Ultralyd i Evaluering av Pasienter Med Mistenkt COVID-19 Infeksjon i Norge
Brief Title: Ultrasonography in Norwegian Emergency Department Patients With Suspected Covid-19 Infection
Acronym: COVIDUS-NOR
Status: Terminated | Type: Observational
Why Stopped: lack of Covid-19 patients
Sponsor: St. Olavs Hospital (Other)
Collaborators: Haukeland University Hospital (Other); Ullevaal University Hospital (Other); Nordlandssykehuset HF (Other); Sorlandet Hospital HF (Other Government); Drammen sykehus (Other); Sykehuset Telemark (Other Government); Helse Stavanger HF (Other Government); University Hospital, Akershus (Other)
Responsible Party: Sponsor
Other Study IDs: REK129805
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: COVID-19; Pneumonia, Viral; Pulmonary Infection
Keywords: Ultrasonography; Norway; Emergency Department; Emergency Physicians
MeSH Terms: conditions — COVID-19; Pneumonia, Viral; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19 suspected: Emergency department patients with suspected or diagnosed COVID-19 disease. All patients will be screened at triage and put into isolation if suspected disease. Ultrasound of the patients lungs will be performed after patient consent and findings will be recorded and categorized (Soldati et al., 2020). The use of ultrasound and registration of data will not affect the regular patient evaluation, treatment or logistics.
  Interventions: Diagnostic Test: Lung ultrasound

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — After verbal consent the enrolled patients' lungs are evaluated with ultrasound while in isolation. The lungs are divided into 3 fields and findings are categorized according to Soldati et al., 2020.
  Other Names: Ultrasonography of the lungs

SUMMARY:
In light of the ongoing COVID-19 epidemic in Norway, it is paramount to develop and utilize clinical tools for assessing and risk stratifying patients with suspected coronary infection in the emergency departments. Diagnostic use of ultrasound in viral pneumonias, including COVID-19 has proved to be very useful. The use of ultrasound will assist in quick detection of lung pathology compatible with increasing severity of the COVID-19 disease. At the same time, the use of ultrasound diagnostics in the emergency department could improve logistics and reduce potential exposure of the corona virus to other health personnel.

The purpose of the study is to assess whether ultrasound findings correlates with physical examination, labs, and other imaging diagnostics in patients with suspected or diagnosed COVID-19 disease, as well as assessing whether ultrasound diagnostics can assist in risk stratification. The project is conducted as a prospective multicenter study where ultrasound diagnostics will be performed on patients with suspected coronary infection in the emergency departments. Data collection takes place as part of the daily clinical evaluation of acute patients in the emergency departments. The project is planned to be completed towards the end of 2025.

ELIGIBILITY:
Inclusion Criteria:

- All emergency department patients with suspected or diagnosed COVID-19.

Exclusion Criteria:

* Negative screening for COVID-19
* recent negative COVID-19 test
* no indication for isolation in the Emergency Department

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pasients referred to the ED with signs and symptoms suspected of COVID-19 (including cough, dyspnea, fever), patient already diagnosed with COVID-19, and patients with risk of being in contact with corona virus will be eligible for study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Mortality | up to 30 days
  30-day mortality
Level-of-care | up to 7 days
  In-hospital treatment level, e.g. discharge from ED, observational unit, ward, ICU.

SECONDARY OUTCOMES:
In-hospital length of stay | Up to 30 days
  in days
Oxygen usage in the emergency department | Within 24 hours
Emergency department length of stay | Within 24 hours
  in hours
Antibiotics usage | Within 24 hours

OTHER OUTCOMES:
Clinical correlation | Within 3 days
  Clinical correlation between ultrasound findings and vital signs, labs, blood gas and other diagnostic modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Petter Bjørnsen, MD, PhD, Principal Investigator — NTNU/St. Olav's Hospital
Locations (9):
- Norway (9):
  - Haukeland universitetssykehus, Bergen
  - Nordland Hospital, Bodø
  - Drammen sykehus, Drammen
  - Sørlandet sykehus, Kristiansand, Kristiansand
  - Akershus University Hospital, Oslo
  - Ullevål University Hospital, Oslo
  - Sykehuset Telemark HF, Skien
  - Stavanger Universitetssjukehus, Stavanger
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No